CLINICAL TRIAL: NCT00971165
Title: A Comparison Between Diuretics and Angiotensin-receptor Blocker Agents in Patients With Stage I Hypertension: PREVER-treatment Study
Brief Title: Diuretics and Angiotensin-Receptor Blocker Agents in Patients With Stage I Hypertension
Acronym: PREVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Flávio Danni Fuchs, Dr., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPPG08621-2
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Hypertension; Cardiovascular Disease
Keywords: Hypertension; Chlorthalidone; Amiloride; Losartan; treatment
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Losartan; Chlorthalidone; Amiloride; Diuretics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorthalidone plus amiloride (Active Comparator): Oral Chlorthalidone plus amiloride up to 25 e 5 mg daily for 18 months
  Interventions: Drug: Chlorthalidone plus amiloride
- losartan (Experimental): Oral losartan up to 100 mg daily, once a day, for 18 month
  Interventions: Drug: losartan

INTERVENTIONS:
Drug: losartan — Oral losartan up to 100 mg daily fo 18 months
  Arms: losartan
Drug: Chlorthalidone plus amiloride — Oral Chlorthalidone plus amiloride up to 25 e 5 mg daily, once a day for 18 months
  Other Names: diuretics
  Arms: Chlorthalidone plus amiloride

SUMMARY:
High blood pressure is the major risk factor for Cardiovascular disease (CVD). The prevalence of hypertension in Brazil was established in population-based studies conducted in different cities and States, varying from 22.3 to 44% of adults.

The benefit of drug treatment of hypertension to prevent major cardiovascular events was consistently demonstrated in a large series of clinical trials controlled by placebo.

Diuretics are at least as efficacious as other blood pressure-lowering drugs, are well tolerated, have longer duration of action and the advantage of very low cost to be used in a population intervention. Chlorthalidone is the more efficacious agent. Its main limitation is to induce hypokalemia in a proportion of patients, an adverse effect that can be antagonized by a potassium-sparing diuretic, as amiloride.

A study comparing diuretic with an ARB agent is therefore recommendable in Brazil, in order to support the decisions of the Health Secretary in regard to blood pressure agents supply for the Brazilian population. Such a study was demanded and funded by the Health and Technology Ministries in Brazil.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is already the leading cause of death in Brazil. The superiority of any particular agent among the groups of blood pressure-lowering drugs was investigated in various clinical trials. ALLHAT, the largest and better designed trial showed that chlorthalidone had similar efficacy to prevent fatal and non-fatal coronary events as an ACE inhibitor (lisinopril) and a calcium channel blocker agent (amlodipine). Chlorthalidone was superior to the other agents in the prevention of other cardiovascular outcomes, particularly heart failure. Amlodipine was superior to valsartan, an angiotensin-receptor blocker (ARB) agent, in the prevention of CHD and stroke. There is no head-to-head comparison between diuretics and ARB agents in the prevention of hard cardiovascular outcomes, and even the comparison of their blood pressure-lowering effects is scarcely described in the literature. Despite this, ARB agents are the leading brands in terms of profits in various countries in the world, including Brazil. This leadership is based on a strong commercial strategy, which includes the distortion of the evidences of clinical trials in favor of these drugs. The idea that they have blood pressure-independent effects is accepted by most, despite the evidences of better designed trials. The option by an ARB agent instead of a diuretic as the first line option in the public health system in Brazil would result in a large expenditure of resources, and there is a pressure to include them in the list of essential drugs provided by the government.

This is a nation-based trial, with 24 clinical centers distributed in 9 States. A Coordinating Committee is responsible for the elaboration of this proposal and for the main decisions of the trial. The organizational chart of the study will include an executive Committee, a safety committee, outcome committee, lab and EKG centers, and the research units.

Research questions

1. Is losartan more efficacious and safe than the association of chlorthalidone with amiloride as the first option to control blood pressure in patients with stage I hypertension?
2. Is losartan more efficacious than the association of chlorthalidone with amiloride as the first option to prevent the development of target-organ damage in patients with stage I hypertension?
3. Is losartan more efficacious than the association of chlorthalidone with amiloride as the first option to prevent the occurrence of major cardiovascular events in patients with stage I hypertension?

Methods

Design: randomized, double-blind, clinical trial, controlled by an active treatment.

Eligible participants: patients older than 40 years of age with Stage I hypertension.

Exclusion criteria: low life expectancy, other indications for the use of diuretics, such as cardiovascular disease, intolerance to the study drugs, pregnancy.

Random allocation: by a computer generated list, stratified by center.

Interventions: Chlorthalidone plus amiloride up to 25 e 5 mg daily, versus losartan up to 100 mg daily. Amlodipine up to 10 mg daily and propranolol up to 160 mg/dia, in an open fashion, will be added if blood pressure is not controlled.

Outcomes:

Primary:

1. Blood pressure variation and proportion of use of add-on drugs.
2. Adverse events.
3. Development or worsening of microalbuminuria and of left ventricular hypertrophy in the EKG.

Secondary: fatal or major cardiovascular events: myocardial infarction, stroke, coronary interventions, heart failure, duplication of creatinine.

Follow-up and duration of the study: consultations for evaluation and enrollment and thereafter consultations at the 3th., 6th., 9th, 12th. and 18th. months.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 40 years of age with stage I hypertension

Exclusion Criteria:

* low life expectancy
* other indications for the use of diuretics, such as cardiovascular disease
* intolerance to the study drugs
* pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2010-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure variation and proportion of use of add-on drugs | 18 months
Adverse events | 18 months
Development or worsening of microalbuminuria and of left ventricular hypertrophy in the EKG. | 18 monyhs

SECONDARY OUTCOMES:
fatal or major cardiovascular events: myocardial infarction, stroke, coronary interventions, heart failure, duplication of creatinine | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Flávio D Fuchs, MD, PhD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Fuchs FD, Fuchs SC, Moreira LB, Gus M, Nobrega AC, Poli-de-Figueiredo CE, Mion D, Bortolotto L, Consolim-Colombo F, Nobre F, Coelho EB, Vilela-Martin JF, Moreno H Jr, Cesarino EJ, Franco R, Brandao AA, de Sousa MR, Ribeiro AL, Jardim PC, Afiune Neto A, Scala LC, Mota M, Chaves H, Alves JG, Sobral Filho DC, Pereira e Silva R, Figueiredo Neto JA, Irigoyen MC, Castro I, Steffens AA, Schlatter R, de Mello RB, Mosele F, Ghizzoni F, Berwanger O. A comparison between diuretics and angiotensin-receptor blocker agents in patients with stage I hypertension (PREVER-treatment trial): study protocol for a randomized double-blind controlled trial. Trials. 2011 Feb 24;12:53. doi: 10.1186/1745-6215-12-53. PMID 21349192
- [Derived] Fuchs FD, Scala LCN, Vilela-Martin JF, Whelton PK, Poli-de-Figueiredo CE, Pereira E Silva R, Gus M, Bortolotto LA, Consolim-Colombo FM, Schlatter RP, Cesarino JE, Castro I, Figueiredo Neto JA, Chaves H, Steffens AA, Alves JG, Brandao AA, de Sousa MR, Jardim PC, Moreira LB, Franco RS, Gomes MM, Afiune Neto A, Fuchs FC, Sobral Filho DC, Nobrega AC, Nobre F, Berwanger O, Fuchs SC. Effectiveness of chlorthalidone/amiloride versus losartan in patients with stage I hypertension and diabetes mellitus: results from the PREVER-treatment randomized controlled trial. Acta Diabetol. 2021 Feb;58(2):215-220. doi: 10.1007/s00592-020-01611-8. Epub 2020 Oct 13. PMID 33047257
- [Derived] Fuchs FD, Scala LC, Vilela-Martin JF, de Mello RB, Mosele F, Whelton PK, Poli-de-Figueiredo CE, de Alencastro PR, E Silva RP, Gus M, Bortolotto LA, Schlatter R, Cesarino EJ, Castro I, Neto JA, Chaves H, Steffens AA, Alves JG, Brandao AA, de Sousa MR, Jardim PC, Moreira LB, Franco RS, Gomes MM, Neto AA, Fuchs FC, Filho DC, Nobrega AC, Nobre F, Berwanger O, Fuchs SC. Effectiveness of chlorthalidone/amiloride versus losartan in patients with stage I hypertension: results from the PREVER-treatment randomized trial. J Hypertens. 2016 Apr;34(4):798-806. doi: 10.1097/HJH.0000000000000837. PMID 26938814